CLINICAL TRIAL: NCT05517733
Title: ASSESSMENT OF SOFT TISSUE HEALING OVER IMMEDIATELY PLACED IMPLANT SEALED WITH PLATELETS RICH FIBRIN (PRF) VERSUS DIODE LASER (A RANDOMIZED CONTROLLED CLINICAL TRIAL)
Brief Title: ASSESSMENT OF SOFT TISSUE HEALING OVER IMMEDIATELY PLACED IMPLANT SEALED WITH PLATELETS RICH FIBRIN (PRF) VERSUS DIODE LASER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nourhan M.Aly (Other)
Responsible Party: Sponsor-Investigator, Nourhan M.Aly, Assistant Lecturer of Dental Public Health, University of Alexandria
Organization: University of Alexandria (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11
Record Dates: First submitted 2022-08-24; First posted 2022-08-26 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Immediate Implant Soft Tissue Healing
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Fibrin (PRF) (Experimental)
  Interventions: Biological: Platelet Rich Fibrin
- Diode laser (Experimental)
  Interventions: Device: Diode laser

INTERVENTIONS:
Biological: Platelet Rich Fibrin — for the preparation of PRF, A well-trained professional nurse drew 10ml of patient blood from the antecubital vein and transferred it to a test tube without anticoagulant. The blood sample was immediately centrifuged for 10-12 minutes at 3000 rpm. L-PRF was ready to use after centrifugation.
  PRF membrane was put over the implant and slightly tucked under the soft tissue periphery, then held in place with a figure-of-8 suture by 0.5 proline suture
  Other Names: PRF
  Arms: Platelet Rich Fibrin (PRF)
Device: Diode laser — * A 980 nm diode laser device (BIOLASE) was applied in a circular motion to the blood formed at the socket orifice at a power of 1W for 1 minute with a continuous wave mode, the application was done without touching the pooling blood and with a non-activated tip of the fiber optic.
  * The laser application cycle was repeated 3-5 times to yield a stable fixed blood clot covering the dental implant with no oozing blood from its periphery.
  Arms: Diode laser

SUMMARY:
Aim of the current study was to assess the efficacy of PRF in comparison to diode laser to promote tissue healing and soft tissue quality after placement of immediate implants.

ELIGIBILITY:
Inclusion Criteria:

* Any non-restorable hopeless tooth: a badly decayed tooth that cannot be restored, tooth with failed endodontic treatment, and teeth with longitudinal fracture.
* Post-extraction sockets type 1 with all bony walls intact; Type I extraction sockets according to Elian classification in 2007 have an intact labial plate of the bone and no soft tissue recession. Therefore, it does not require a mucoperiosteal flap elevation, only bone graft particles are packed into the socket after atraumatic extraction and socket debridement, then sealed with barrier membranes or soft tissue grafts.
* No signs of active periodontal disease in the selected tooth.
* Good oral hygiene

Exclusion Criteria:

* The presence of any systemic disease could complicate bone or soft tissue healing after immediate implant placement.
* The presence of Acute periapical infection.
* The presence of any local factor that may interfere with extraction as tooth ankyloses
* Subjects who had undergone therapeutical radiation. (187)
* Patients who had been subjected to or who were under bisphosphonate therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Soft tissue healing | up to 4 weeks
  This was done using Landry healing index. It evaluates the parameters of tissue colour, bleeding response to palpation, presence of granulation tissue, characteristics of the incision margins, and the presence of suppuration. The score ranges from 1 (Very poor) to 5 (Excellent).
Mid-buccal soft tissue thickness | up to 8 weeks
  Measured from the gingival margin to implant platform using a periodontal probe.
Mid-crestal soft tissue height | up to 8 weeks
  Measured using a periodontal probe passing through soft tissue in the intersection midpoint of both buccolingual and mesiodistal dimensions of the socket till cover screw.

SECONDARY OUTCOMES:
Post-operative pain level | 24 hours
  This was measured using the Visual Analogue Scale (VAS) that rates pain level on a scale of 0-10 (with 0 meaning no pain at all and 100 meaning the worst possible pain). A VAS questionnaire was given to the subjects and they were asked to select their pain score.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt